CLINICAL TRIAL: NCT00004296
Title: Multicenter Study of Nontuberculous Mycobacteria in Cystic Fibrosis Patients
Status: Completed | Type: Observational
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: University of North Carolina (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Other Study IDs: 199/11731; UNCCH-939
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2000-01

CONDITIONS: Cystic Fibrosis; Atypical Mycobacterium Infection
Keywords: atypical mycobacterium infection; bacterial infection; cardiovascular and respiratory diseases; cystic fibrosis; genetic diseases and dysmorphic syndromes; immunologic disorders and infectious disorders; mycobacterium infection; rare disease
MeSH Terms: conditions — Cystic Fibrosis; Mycobacterium Infections, Nontuberculous; Bacterial Infections; Respiratory Tract Diseases; Genetic Diseases, Inborn; Immune System Diseases; Communicable Diseases; Mycobacterium Infections; Rare Diseases

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
OBJECTIVES: I. Determine the prevalence of nontuberculous mycobacteria in sputum cultures from patients with cystic fibrosis.

II. Compare the clinical course of patients with negative versus positive cultures.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Participants are screened for nontuberculous mycobacteria (NTM) with 3 sputum acid-fast bacilli smears and mycobacterial cultures, with speciation of positive cultures, collected over 1 year. Demographic data, diagnostic criteria, clinical measurements, and other respiratory pathogen data are collected using the Cystic Fibrosis Foundation Patient Registry Questionnaire.

NTM-positive patients (cases) matched with NTM-negative controls identified in screening are followed every 3 months for 15 months. Cases are evaluated for NTM burden during the first 3 months.

Appropriate therapy is offered to consistently NTM-positive cases. Lung transplant recipients are removed from study.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

Patients over age 10 with cystic fibrosis documented as follows:

* Pilocarpine sweat chloride test at least 60 mEq/L OR
* Genotyping or transepithelial potential difference AND
* Clinical symptoms of suppurative respiratory disease or pancreatic insufficiency

Able to produce at least 3 sputum samples

* Bronchoscopy specimens acceptable
* Throat/nasal specimens not acceptable

No Pseudomonas cepacia colonization

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000
Dates: Start 1995-09

CONTACTS AND LOCATIONS:
Overall Officials: Ken Olivier, Study Chair — University of North Carolina

REFERENCES:
- [Background] Whittier S, Olivier K, Gilligan P, Knowles M, Della-Latta P. Proficiency testing of clinical microbiology laboratories using modified decontamination procedures for detection of nontuberculous mycobacteria in sputum samples from cystic fibrosis patients. The Nontuberculous Mycobacteria in Cystic Fibrosis Study Group. J Clin Microbiol. 1997 Oct;35(10):2706-8. doi: 10.1128/jcm.35.10.2706-2708.1997. PMID 9316943
- [Background] Olivier KN.: Collaborative CFF/NCRR study of the epidemiology of nontuberculous mycobacteria in cystic fibrosis. Pediatric Pulmonology Suppl. 19: 145-146, 1999.